CLINICAL TRIAL: NCT06673095
Title: ICEMAN (Intelligent Choice of Excision Margin): A Randomized Controlled Trial of Narrow Excision Versus Wide Excision for Adults With Primary Invasive Cutaneous Melanomas
Brief Title: Narrow Excision Versus Wide Excision for the Treatment of Adults With Invasive Cutaneous Melanoma, ICEMAN Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Wesley Yu, M.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00027175; NCI-2024-08327 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00027175 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-10-22; First posted 2024-11-04 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Clinical Stage IA Cutaneous Melanoma AJCC v8; Clinical Stage IB Cutaneous Melanoma AJCC v8
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (narrow margin excision) (Experimental): Patients undergo narrow margin excision on study. Patients may optionally undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Excision; Other: Survey Administration
- Arm II (wide margin excision) (Active Comparator): Patients undergo wide margin excision on study. Patients may optionally undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Excision; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Excision — Undergo narrow margin excision
  Other Names: Abscission; Extirpation; Surgical Removal
  Arms: Arm I (narrow margin excision)
Procedure: Excision — Undergo wide margin excision
  Other Names: Abscission; Extirpation; Surgical Removal
  Arms: Arm II (wide margin excision)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial compares the effect of a narrow surgical excision (removal) to a wide excision for the treatment of adults with invasive cutaneous melanoma. Currently the standard of care is to take wide margins (boarder of healthy tissue surrounding the melanoma) when removing melanoma. Narrow margin excision removes a smaller amount of healthy tissue when surgically removing the melanoma. Narrow margin excision may be effective in removing the melanoma while also reducing surgical complications and improving quality of life for adults with invasive cutaneous melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the 3-year local recurrence-free survival rates (RFS) in melanoma patients treated with narrow excision versus (vs) wide excision.

SECONDARY OBJECTIVES:

I. To measure the 3-, 5-year Regional (nodal) disease-free survival (DFS) in melanoma patients treated with active nodal surveillance.

II. To compare 5-year local recurrence-free survival in patients treated with narrow vs wide excision.

III. To compare 5-year Melanoma Specific Survival (MSS) in patients treated with narrow vs wide excision.

IV. To compare the quality of life in patients treated with narrow vs wide excision.

V. To compare surgical complication rates in patients treated with narrow vs wide excision.

VI. To compare the frequency of complex reconstruction in patients treated with narrow vs wide excision.

VII. To compare the final defect size in patients treated with narrow vs wide excision.

VIII. To compare the number of operative/procedure days required to achieve negative margins.

EXPLORATORY OBJECTIVE:

I. To measure the T- and B-cell repertoires in patients with melanoma over time.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo narrow margin excision on study. Patients may optionally undergo blood sample collection throughout the study.

ARM II: Patients undergo wide margin excision on study. Patients may optionally undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 1 week, 3, 6, 12, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants or legally authorized representatives (LAR) must provide written informed consent before any study-specific procedures or interventions are performed
* Age ≥ 18 years; all biological gender identities and racial/ethnic groups will be included
* Participants must have histologically confirmed primary cutaneous melanoma. Acral melanomas are eligible.
* Participants must have one of the following:

  * American Joint Committee on Cancer (AJCC) 8th Ed clinical stage IA disease with Breslow thickness ≥ 0.5 mm AND at least one high-risk feature (Mitotic rate ≥ 2/mm2, age ≤ 42, lymphovascular invasion, head/neck location)
  * AJCC 8th Ed Clinical Stage IB melanoma

    * If a melanoma is widely transected and the true Breslow depth is uncertain, then to be eligible for this trial, the melanoma must be re-biopsied to ascertain an accurate Breslow depth.
* The index melanoma must be classified as low risk on the Merlin Assay (SkylineDx)
* Study intervention (surgery) must be completed within 120 days of the original diagnostic biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 50%)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants with a history of HIV infection are eligible
* Participants can speak, read and write in English or Spanish

Exclusion Criteria:

* Uncertain diagnosis of melanoma (i.e. severely dysplastic nevi, melanocytic lesion of unknown malignant potential, atypical intraepidermal melanocytic proliferations)
* The patient has already undergone wide local excision at the site of the primary index lesion
* The patient has a pure desmoplastic melanoma. A pure desmoplastic melanoma is defined as being > 90% desmoplastic type. Melanomas with < 90% desmoplastic type may be included in this trial
* Mucosal and ocular melanomas are also excluded, as these are approached differently for surgical excision
* Physical, clinical, radiographic, or pathologic evidence of satellite, in-transit, regional, or distant metastatic melanoma
* Participants with known or suspected cancer with regional or distant metastasis are excluded from this clinical trial because this trial is aimed at evaluating the control of localized disease
* The patient has undergone surgery on a separate occasion to clear the lymph nodes of the probable draining lymphatic field, including a sentinel lymph node biopsy, of the index melanoma
* Planned adjuvant radiotherapy to the primary melanoma site after excision
* Participant is unwilling or unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Local recurrence rate | From randomization to end of year 3
  Defined as average rate at which cancer returns to same location as the original tumor.

SECONDARY OUTCOMES:
Regional (nodal) disease-free survival | From randomization to end of year 5
  Average number of participants who are experiencing regional disease-free survival at 3 and 5 years.
Local recurrence-free survival | From randomization to end of year 5
  The average length of time (in months) from the date of randomization to local recurrence.
Melanoma-specific survival | From randomization to end of year 5
  The average length of time (in months) from date of randomization to death.
Postoperative pain | Up to 30 days after surgery
  Measured by numeric rating scale (0-10).
Quality of life | Up to postoperative day 90
  Quality of life score as measured by either the Facial Appearance, Quality of Life, and Experience Questionnaire (FACE-Q) score in patients with melanoma on the face or the Functional Assessment of Cancer Therapy - Melanoma (FACT-M) score for patients with melanoma elsewhere on the body. FACT-M is a tool for measuring health-related quality of life in patients with melanoma. It has 51 items, Scores range from 0 to 120 with higher score indicating better quality of life (QOL). FACE-Q includes 5 independently functioning scales and 2 checklists that measure outcomes important to patients from their perspective.
Surgical complication rate | Up to postoperative day 90
  Defined as the proportion of patients experiencing a surgical complication.
Frequency of complex reconstruction | Immediately after surgery
  Defined as the proportion of patients receiving any flap or graft reconstruction.
Defect size | Immediately after surgery
  The size of the defect is measured as the greatest dimension of the final wound multiplied by the dimension perpendicular to the greatest dimension.
Number of operative/procedure days | Up to postoperative day 90
  Will compare the number of operative/procedure days required to achieve negative margins. Will be reported and compared separately (Mohs surgery, narrow excision with permanent sections, wide excision with permanent sections, and slow Mohs).

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Yu, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Bichakjian CK, Swetter SM, Carroll BT, Vidal NY, Simons EA, Vetto JT, Yu WY. ICEMAN (Intelligent Choice of Excision Margin): A Randomized Controlled Trial of Adaptive Narrow Excision Versus Wide Excision for Adults with AJCC Stage I Cutaneous Melanoma. Ann Surg Oncol. 2025 Dec;32(13):9488-9490. doi: 10.1245/s10434-025-18282-w. Epub 2025 Sep 8. PMID 40921901